CLINICAL TRIAL: NCT03313258
Title: The Relationship Between the Use of a Continuous a Zero-heat Flux Temperature Monitor on Initial Discharge Hypothermia Rate Among Severely Injured Trauma Patients: a Randomized Controlled Trial. (RUZIT Trial)
Brief Title: Zero Heat Flux Temp Monitor on Discharge Hypothermia Among Trauma Patients (RUZIT Trial)
Acronym: RUZIT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Dr. Asim Alam (Other)
Responsible Party: Sponsor-Investigator, Dr. Asim Alam, MD, FRCPC, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: RUZIT
Record Dates: First submitted 2017-10-04; First posted 2017-10-18 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Hypothermia; Trauma; Temperature Change, Body
MeSH Terms: conditions — Hypothermia; Wounds and Injuries; Body Temperature Changes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Group (Active Comparator): ZHF temperature monitor cable will be placed appropriately on the forehead by the care team under the direction of the research personnel. The research personnel will then connect this cable to a screen that is blinded to the care team but not to the research personnel.
  Interventions: Device: Standard of Care Group
- Active Warming Group (Experimental): ZHF temperature monitor cable will be placed appropriately on the forehead by the care team under the direction of the research personnel. The research personnel will then connect this cable to a screen that is un-blinded to everyone so healthcare practitioners will be able to visually detect continuous temperature readings from the ZHF monitor.
  Interventions: Device: Active Warming Group

INTERVENTIONS:
Device: Standard of Care Group — ZHF temperature monitor cable will be placed appropriately on the forehead by the care team under the direction of the research personnel. The research personnel will then connect this cable to a screen that is blinded to the care team but not to the research personnel.
  Arms: Standard of Care Group
Device: Active Warming Group — ZHF temperature monitor cable will be placed appropriately on the forehead by the care team under the direction of the research personnel. The research personnel will then connect this cable to a screen that is un-blinded to everyone so healthcare practitioners will be able to visually detect continuous temperature readings from the ZHF monitor.
  Arms: Active Warming Group

SUMMARY:
Hypothermia amongst trauma patients is a persistent problem that increases the relative risk of transfusion as well as morbidity and mortality. The investigators propose to conduct a single-centered randomized controlled trial to determine if the use of a zero-heat flux (ZHF) temperature monitor can reduce the incidence of hypothermia amongst trauma patients discharged from the trauma bay (TB). All eligible trauma patients will be randomized to either a standard of care group or an active temperature monitoring group. In the active temperature monitoring group, a ZHF monitor will be placed on respective trauma patients to continuously record their temperatures after they enter the TB at a large tertiary trauma centre, Sunnybrook Health Sciences Centre (SHSC), in Toronto, ON. The investigators will determine if early continuous temperature monitoring can reduce the incidence of hypothermia upon discharge from the TB. Should early monitoring of severely injured trauma patients within the hospital improves discharge temperature, the foundation for two additional research studies will be laid. Firstly, the investigators will enter a vanguard phase of this trial and assess if early warming patients can improve morbidity and mortality in this patient population utilizing a multi-centered randomized controlled trial design. This will be further extended to test whether early monitoring can be applied in a pre-hospital setting (i.e. within ambulances and transport vehicles) to improve admission temperatures in the TB.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Severely injured trauma patients with a Revised Trauma Score (RTS) ≤ 11 brought into the SHSC TB.

Exclusion Criteria:

* Patients with blast injuries to the face or severe facial trauma will be excluded.
* Major burn patients - as they follow a separate care pathway at SHSC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Hypothermic (<36°C) upon discharge from the trauma bay | Duration of their stay in the trauma bay or up to 4 hours in the trauma bay (whichever comes first)
  Proportion of patients who are hypothermic (<36°C) upon discharge from the trauma bay.

SECONDARY OUTCOMES:
Warming initiatives | Duration of their stay in the trauma bay or up to 4 hours in the trauma bay (whichever comes first)
  Total number of warming initiatives implemented by trauma care team
Transfused products | Duration of their stay in the trauma bay or up to 4 hours in the trauma bay (whichever comes first)
  Number of transfused blood products
Length of stay | Time of admission to discharge or up to 1 year after admission (whichever comes first)
  Number of days patient stayed in hospital
30 day mortality | Time of admission to discharge or up to 30 days after admission (whichever comes first)
  Alive or deceased at 30 day

CONTACTS AND LOCATIONS:
Overall Officials: Asim Alam, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jurkovich GJ, Greiser WB, Luterman A, Curreri PW. Hypothermia in trauma victims: an ominous predictor of survival. J Trauma. 1987 Sep;27(9):1019-24. PMID 3656464
- [Background] Luna GK, Maier RV, Pavlin EG, Anardi D, Copass MK, Oreskovich MR. Incidence and effect of hypothermia in seriously injured patients. J Trauma. 1987 Sep;27(9):1014-8. doi: 10.1097/00005373-198709000-00010. PMID 3656463
- [Background] Wang HE, Callaway CW, Peitzman AB, Tisherman SA. Admission hypothermia and outcome after major trauma. Crit Care Med. 2005 Jun;33(6):1296-301. doi: 10.1097/01.ccm.0000165965.31895.80. PMID 15942347
- [Background] Shafi S, Elliott AC, Gentilello L. Is hypothermia simply a marker of shock and injury severity or an independent risk factor for mortality in trauma patients? Analysis of a large national trauma registry. J Trauma. 2005 Nov;59(5):1081-5. doi: 10.1097/01.ta.0000188647.03665.fd. PMID 16385283
- [Background] Perlman R, Callum J, Laflamme C, Tien H, Nascimento B, Beckett A, Alam A. A recommended early goal-directed management guideline for the prevention of hypothermia-related transfusion, morbidity, and mortality in severely injured trauma patients. Crit Care. 2016 Apr 20;20(1):107. doi: 10.1186/s13054-016-1271-z. PMID 27095272
- [Background] Bukur M, Hadjibashi AA, Ley EJ, Malinoski D, Singer M, Barmparas G, Margulies D, Salim A. Impact of prehospital hypothermia on transfusion requirements and outcomes. J Trauma Acute Care Surg. 2012 Nov;73(5):1195-201. doi: 10.1097/TA.0b013e31826fc7d9. PMID 23117380
- [Background] Rajagopalan S, Mascha E, Na J, Sessler DI. The effects of mild perioperative hypothermia on blood loss and transfusion requirement. Anesthesiology. 2008 Jan;108(1):71-7. doi: 10.1097/01.anes.0000296719.73450.52. PMID 18156884
- [Background] Sun Z, Honar H, Sessler DI, Dalton JE, Yang D, Panjasawatwong K, Deroee AF, Salmasi V, Saager L, Kurz A. Intraoperative core temperature patterns, transfusion requirement, and hospital duration in patients warmed with forced air. Anesthesiology. 2015 Feb;122(2):276-85. doi: 10.1097/ALN.0000000000000551. PMID 25603202
- [Background] Malone DL, Dunne J, Tracy JK, Putnam AT, Scalea TM, Napolitano LM. Blood transfusion, independent of shock severity, is associated with worse outcome in trauma. J Trauma. 2003 May;54(5):898-905; discussion 905-7. doi: 10.1097/01.TA.0000060261.10597.5C. PMID 12777902
- [Background] Bochicchio GV, Napolitano L, Joshi M, Bochicchio K, Meyer W, Scalea TM. Outcome analysis of blood product transfusion in trauma patients: a prospective, risk-adjusted study. World J Surg. 2008 Oct;32(10):2185-9. doi: 10.1007/s00268-008-9655-0. PMID 18575931
- [Background] Perel P, Clayton T, Altman DG, Croft P, Douglas I, Hemingway H, Hingorani A, Morley KI, Riley R, Timmis A, Van der Windt D, Roberts I; PROGRESS Partnership. Red blood cell transfusion and mortality in trauma patients: risk-stratified analysis of an observational study. PLoS Med. 2014 Jun 17;11(6):e1001664. doi: 10.1371/journal.pmed.1001664. eCollection 2014 Jun. PMID 24937305
- [Background] Dunne JR, Riddle MS, Danko J, Hayden R, Petersen K. Blood transfusion is associated with infection and increased resource utilization in combat casualties. Am Surg. 2006 Jul;72(7):619-25; discussion 625-6. PMID 16875084
- [Background] Bochicchio GV, Napolitano L, Joshi M, Bochicchio K, Shih D, Meyer W, Scalea TM. Blood product transfusion and ventilator-associated pneumonia in trauma patients. Surg Infect (Larchmt). 2008 Aug;9(4):415-22. doi: 10.1089/sur.2006.069. PMID 18759678
- [Background] Reynolds BR, Forsythe RM, Harbrecht BG, Cuschieri J, Minei JP, Maier RV, Moore EE, Billiar EE, Peitzman AB, Sperry JL; Inflammation and Host Response to Injury Investigators. Hypothermia in massive transfusion: have we been paying enough attention to it? J Trauma Acute Care Surg. 2012 Aug;73(2):486-91. PMID 23019675
- [Background] Lapostolle F, Sebbah JL, Couvreur J, Koch FX, Savary D, Tazarourte K, Egman G, Mzabi L, Galinski M, Adnet F. Risk factors for onset of hypothermia in trauma victims: the HypoTraum study. Crit Care. 2012 Jul 31;16(4):R142. doi: 10.1186/cc11449. PMID 22849694
- [Background] Eshraghi Y, Nasr V, Parra-Sanchez I, Van Duren A, Botham M, Santoscoy T, Sessler DI. An evaluation of a zero-heat-flux cutaneous thermometer in cardiac surgical patients. Anesth Analg. 2014 Sep;119(3):543-549. doi: 10.1213/ANE.0000000000000319. PMID 25045862